CLINICAL TRIAL: NCT01146977
Title: Autologous Hematopoietic Cell Transplantation for Core-binding Factor Positive Acute Myeloid Leukemia in the First Complete Remission
Brief Title: Autologous Hematopoietic Cell Transplantation for Core-binding Factor (CBF) Acute Myeloid Leukemia (AML) in the First Complete Remission (CR1)
Acronym: CBF(+)AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: COSAH, Cooperative Study Group A for Hematology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-020
Record Dates: First submitted 2010-05-19; First posted 2010-06-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: CBF(+)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous HCT (Experimental): 5.1.3. After achieving CR1, patient will be invited to this protocol and will be able to decide whether to join or not after listening to the information.
  5.1.3.1. If he/she decides to participate, request of health insurance support on the autologous HCT will be submitted and further processes related to autologous HCT will continue.
  Interventions: Other: Autologous HCT
- HDAC chemotherapy (Active Comparator): If he/she decides not to participate, he/she will be treated with HDAC consolidation chemotherapy, which is the current standard treatment.
  Interventions: Other: HDAC chemotherapy

INTERVENTIONS:
Other: HDAC chemotherapy — If he/she decides not to participate, he/she will be treated with HDAC consolidation chemotherapy, which is the current standard treatment.
  Other Names: Cytarabine 3g/m2
  Arms: HDAC chemotherapy
Other: Autologous HCT — After achieving CR1, patient will be invited to this protocol and will be able to decide whether to join or not after listening to the information.
  If he/she decides to participate, request of health insurance support on the autologous HCT will be submitted and further processes related to autologous HCT will continue.
  Arms: Autologous HCT

SUMMARY:
Evaluation of efficacy of autologous hematopoietic cell transplantation (HCT) with core-binding factor (CBF) positive acute myeloid leukemia (AML) in the first CR (CR1).

DETAILED DESCRIPTION:
5.2 AUTOLOGOUS PBSCS HARVESTING

5.2.1. PBSCs will be collected during recovery phase after the second cycle of HDAC consolidation chemotherapy.

5.2.2. For mobilization, recombinant human granulocyte- colony-stimulating factor (G-CSF, Filgrastim) will be given subcutaneously at a dose of 10 mcg/kg from day 9 of the 2nd HDAC cycle until the completion of harvesting.

5.2.3. PBSCs harvesting will be performed via perm-cath or Quinton catheter, which will be inserted with fluoroscopy-guided before starting and will be removed after finishing harvest.

5.2.4. Harvest will be initiated from the day when the peripheral absolute neutrophil count reach up to 0.2 x 109/mm3. Peripheral blood mononuclear cells will be collected by leukapheresis method with 'CS-3000' (Baxter, Deerfield, IL) or other compatible machine. Cell collection will be performed for at least 2 days and the duration of collection can be extended until a target CD34+ cell dose of 5 x 106/kg (in terms of body weight of recipient) is collected.

5.2.5. If adequate numbers of CD34+ cells are not collected, the 3rd HDAC chemotherapy will be done and mobilization/harvest procedure will be repeated.

5.2.6. Stem cells harvested from patient will be frozen in liquid nitrogen tank for future autologous HCT cell infusion.

5.3.PRETRANSPLANT WORKUP FOR AUTOLOGOUS HCT 5.3.1. Pre-workup for checking the current disease status and feasibility for autologous HCT will be performed before the conditioning and infusion of autologous HCT.

5.3.2. It is recommended that baseline workup for hematologic / non-hematologic status will be performed at least 1 month prior to the initiation of conditioning. Bone marrow aspirate/ biopsy with cytogenetics and diagnostic lumbar puncture can be performed immediately before the initiation of conditioning.

5.3.3. Pretransplant workup tests are listed in Appendix IV.

5.4. CONDITIONING REGIMEN FOR AUTOLOGOUS HCT 5.4.1. On admission, 5.4.1.1.Menstruating women will be given norethindrone (Norlutate) 10mg po daily until platelet count is consistently over 100,000 /mcL.

5.4.1.2.Actual body weight (ABW) for busulfan will be calculated using following guidelines; 5.4.1.2.1.If ABW is less or equal to ideal body weight (IBW), use ABW. 5.4.1.2.2.If ABW is greater than IBW but ABW is within 120% of IBW, use IBW. 5.4.1.2.3.If ABW is 120% or greater than IBW, use IBW+25% (ABW-IBW). 5.4.1.2.4.IBW(ideal body weight) will be calculated in 5.4.1.2.4.1.Male: 50 kg + 2.3kg (height[inch]-60) 5.4.1.2.4.2.Female: 45.5kg + 2.3kg (height[inch]-60) 5.4.1.2.4.3.1inch=2.54cm 5.4.2. On day -8, preparation drugs will be administered to patient as below; 5.4.2.1.Hydration with 0.9% normal saline will be started at 6PM and infused continuously at a rate of 100mL/hr through day -4.

5.4.2.2.Allopurinol 300mg/day will be taken p.o. once a day from day-8 to -2. 5.4.2.3.Heparin 100 U/kg/day in normal saline 500 mL will be infused continuously at a rate of 20mL/hr through day 20 (6pm). Heparin should be discontinued if there is clinically significant bleeding or aPTT level exceeds 1.2 time of the upper normal limit.

5.4.2.4.Dilantin 15mg/kg (ABW) in normal saline 300cc will be infused continuously at a rate of 200mL/hr at 8PM, and then, 200mg will be taken p.o. twice a day through day -4. Dilantin level should be monitored in the morning of day-7 and -6 to maintain the level within 10 to 20 mg/L.

5.4.3. From day-7, conditioning drug will be administered to patient as below; 5.4.3.1.Busulfan 3.2mg/kg/day in normal saline of 10 times the volume of busulfan will be infused continuously over 3 hours with an interval of 24 hours on days -7 to -5 (for 3 days).

5.4.3.2.Etoposide 200mg/m2/day in normal saline 1000mL will be infused continuously over 5 hours twice a day with an interval of 12 hours on day-3 to -2 (for 2 days).

5.4.3.3.Antiemetics such as serotonin antagonist or lorazepam are allowed.

5.5. AUTOLOGOUS PBSCS INFUSION 5.5.1. Autologous PBSCs will be infused on day0. 5.5.1.1.Premedication including pheniramine maleate (avil) 45.5mg i.v., acetaminophen 600mg p.o., hydrocortisone 250mg i.v. and furosemide 20mg i.v. will be given 30 minutes before cell infusion.

5.5.1.2.PBSCs will be infused via saline infusion set without in-line filters. 5.5.1.3.Vital sign should be checked 4 times with 15 minutes of interval, 4 times with 30 minutes, and then 4 times with 1 hour. Electrocardiogram monitoring will be performed from the start until the completion of PBSCs infusion.

5.5.1.4.Following medications should not be administered simultaneously with PBSCs; 5.5.1.4.1.Lipid-containing total parenteral nutrition fluid 5.5.1.4.2.Conventional or liposomal amphotericin 5.6. SUPPORTIVE CARE 5.6.1. Recombinant human G-CSF (rhG-CSF) 450㎍ in 100 mL of D5W will be infused intravenously over 30 minutes from day 5 till ANC>3,000/㎕.

5.6.2. Ciprofloxacin 500mg will be given p.o. twice a day (for selective bowel decontamination) from day 1 till ANC>3,000/㎕. With the first fever spike, ciprofloxacin can be replaced with broad spectrum antibiotics.

5.6.3. Micafungin 50mg will be infused intravenously once a day from day1 till ANC>3,000/㎕.

5.6.4. Acyclovir 250mg/m2 will be infused twice a day from day1 till ANC>3,000/㎕.

5.6.5. In case of oral mucositis, sodium bicarbonate/saline mouthwash will be applied four times a day until resolved.

5.6.6. Clotrimazole or Canesten® powder can be applied to groin, axilla, and perianal area twice a day from day-8 until engraftment.

5.6.7. All cellular blood products must be transfused after leukocyte filtration and irradiation.

5.6.8. For woman of childbearing potential, adequate consultation for ovarian protection can be sought. For man who intend to have child(ren) in future, sperm banking can be recommended and performed.

5.7. EVALUATION DURING TREATMENT 5.7.1. CBC with differential count, ALT/AST, bilirubin with BUN/Cr, and electrolyte will be checked once daily.

5.7.2. Chemical battery with BUN/phosphorus, LDH and level of magnesium will be checked three times a week.

5.7.3. Coagulation battery with fibrinogen/d-dimer will be checked at day 0, 7, 14, 21 and once a week thereafter until discharge.

5.7.4. Protein C, antithrombin III, t-PA antigen, and PAI-1 antigen will be checked at day 0, 7, 14, and 21.

5.7.5. Urinalysis will be checked once a week. 5.7.6. Chest X-ray will be checked once a week routinely and more frequently according to patient's condition.

5.7.7. Blood galactomannan (aspergillosis antigen, GM) assay can be recommended to be checked once a week until ANC>3,000/ according to the physician's decision.

5.8. POST-HCT FOLLOW-UP INCLUDING MRD MONITORING 5.8.1. Patients will be followed with physical examination and appropriate blood test including CBC at least every 3 months for 3 years, every 6 months for the next 2 years, and then annually thereafter.

5.8.2. Toxicities related to treatment will be assessed and reported according to NCI CTCAE v3.0.

5.8.3. Minimal residual disease (MRD) monitoring with RQ-PCR for AML1/ETO or CBFβ/MYH11 will be performed before autologous HCT (bone marrow and peripheral blood, 1 month after autologous HCT (bone marrow and peripheral blood), and thereafter, every 3 months (peripheral blood only) until 3 years after autologous HCT.

5.8.4. If RQ-PCR is not available, RT-PCR and/or FISH can be used for MRD monitoring

ELIGIBILITY:
Inclusion Criteria:

* Patients with CBF positive AML in CR1. CBF AML includes t(8;21)(q22;q22) [AML1(RUNX1)/ETO(CBFα2T1)], inv(16)(q13q22) (CBFβ/MYH11),t(16;16)(p13;q22) (CBFβ/MYH11) Using RT-PCR, FISH, or standard karyotype analysis technique.
* Patients who plan to receive the second cycle of HDAC consolidation chemotherapy.
* 15 years old or older and 65 years or younger
* Adequate performance status (Karnofsky score of 70 or more).
* Adequate hepatic and renal function (AST, ALT, and bilirubin < 3.0 x upper normal limit, and creatinine < 2.0 mg/dL).
* Adequate cardiac function (left ventricular ejection fraction over 40% on heart scan or echocardiography)
* Signed and dated informed consent must be obtained from patient.

Exclusion Criteria:

* Presence of significant active infection
* Presence of uncontrolled bleeding
* Any coexisting major illness or organ failure
* Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible
* Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-01 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
CIR, DFS | 6 years
  * Relapse incidence (cumulative incidence of relapse, CIR)
  * Disease-free survival (DFS)

SECONDARY OUTCOMES:
TRM, EFS, OS | 6 years
  * Engraftment rate / time to engraftment
  * Transplantation-related mortality (TRM)
  * Event-free survival (EFS)
  * Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Dae-Young Kim, professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Asanbyeongwon-gil, Songpa-gu, South Korea

REFERENCES:
- See also: Autologous hematopoietic cell transplantation for core-binding factor positive acute myeloid leukemia in the first complete remission — http://www.google.co.kr